CLINICAL TRIAL: NCT02182245
Title: A Phase I Open Label Dose Escalation Study of Oral Treatment With BIBF 1120 in Combination With Standard Treatment of Paclitaxel and Carboplatin in Patients With Advanced Gynaecological Malignancies
Brief Title: Dose Escalation Study of BIBF 1120 in Patients With Advanced Gynaecological Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1199.6
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Genital Neoplasms, Female
MeSH Terms: conditions — Genital Neoplasms, Female | interventions — nintedanib; Paclitaxel; Carboplatin

ARMS (2):
- Combination Therapy (Experimental)
  Interventions: Drug: BIBF 1120; Drug: Paclitaxel; Drug: Carboplatin
- Monotherapy (Experimental)
  Interventions: Drug: BIBF 1120

INTERVENTIONS:
Drug: BIBF 1120
Drug: Paclitaxel
  Arms: Combination Therapy
Drug: Carboplatin
  Arms: Combination Therapy

SUMMARY:
The primary objectives of this trial were to determine the safety, tolerability, and MTD of BIBF 1120 when added to standard therapy with carboplatin and paclitaxel

ELIGIBILITY:
Inclusion Criteria:

* Female patients with the following histologically confirmed advanced gynaecological malignancies: epithelial ovarian cancer, endometrial carcinoma, uterine sarcoma, mixed Müllerian tumour, fallopian tube carcinoma, primary peritoneal carcinoma, cervical carcinoma or vulvular carcinoma
* Metastatic disease or locally advanced disease that is not resectable with curative intention
* Indication for combination chemotherapy with paclitaxel/carboplatin as judged by the investigator
* Age 18 years or older
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Life expectancy of at least 6 months
* Written informed consent that is not consistent with ICH-GCP (International Conference on Harmonisation - Good Clinical Practice) guidelines and local requirements

Exclusion Criteria:

* Participation in another clinical study within the past 4 weeks before start of therapy or concomitantly with this study
* Radiotherapy within 4 weeks before the start of therapy
* Chemotherapy, immunotherapy or hormonal therapy (with the exception of hormonal replacement therapy) within 4 weeks before the start of the therapy
* Patients with germ cell tumours, early stage ovarian cancer (Fédération Internationale de Gynécologie et d'Obstétrique [FIGO] stage I-IIA), primary cervical cancer (FIGO I-III), primary endometrial cancer (FIGO I-III) or borderline tumours
* Patients with known brain metastases
* Symptomatic bowel obstruction or known or suspected malabsorption
* Patients with pericardial effusion which is haemodynamically relevant
* Other malignancy diagnosed within the past 5 years (other than non-melanomatous skin cancer or cervical carcinoma in situ)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study medication
* History of haemorrhagic or thrombotic event (including transient ischemic attacks) in the past 6 months
* Concurrent therapeutic anticoagulation or anti-platelet therapy (except chronic low dose daily acetylsalicylic acid <300 mg)
* Major injuries and surgeries within the past 3 weeks, planned surgical procedures during the trial, incomplete wound healing
* Known hypersensitivity to paclitaxel, carboplatin, BIBF 1120 or any of their excipients or vehicles such as polyoxyethylated castor oil
* Clinically significant peripheral polyneuropathy (>CTCAE grade 1) which precludes therapy with paclitaxel
* Absolute neutrophil count (ANC) <1500/μL, platelet count <100000/μL, or haemoglobin <9 mg/dL
* Total bilirubin >1.5 mg/dL (26 μmol/L), ALT (Alanine aminotransferase) and/or AST (Aspartate aminotransferase) >1.5 x the upper limit of normal (ULN)
* Serum creatinine >1.5 mg/dL (>132 μmol/L)
* Persistent gross haematuria
* Pregnancy or breast feeding
* Women with childbearing potential and who are sexually active and unwilling to use a medically acceptable method of contraception (oral contraceptive, diaphragm with spermicide, intrauterine device, condom with spermicide)
* Known or suspected active drug or alcohol abuse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-10-01 (Actual); Primary Completion 2007-01-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of BIBF 1120 | up to 126 days
Incidence and intensity of adverse events according to the CTCAE (Common terminology criteria for adverse events Version) version 3.0 with increasing doses of BIBF 1120 | up to 9 months

SECONDARY OUTCOMES:
Objective tumour response after treatment with BIBF 1120 in combination with carboplatin and paclitaxel in evaluable patients | up to 9 months
Cancer antigen 125 (CA-125) response | Day 1 of each treatment period
Time to tumour progression (time from treatment start to the time of documented tumour progression) | up to 9 months

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com